CLINICAL TRIAL: NCT05342480
Title: Intensive Two Week Inpatient Trauma Treatment. A Pilotstudy.
Brief Title: Intensiv Inpatient Trauma Treatment. A Pilotstudy.
Acronym: ITBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Julie Horgen Evensen, Consultant, Research coordinator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 453358
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Pilot study PTSD trauma treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EMDR and PE combined treatment — Daily program monday to friday with daily PE and EMDR sessions, physical activity between sessions, in vivo exposure treament and psychoeducational groups. Daily rotation of both EMDR and PE therapists. Multidisiplinary team attached to each pati

SUMMARY:
Aim of the study: Post traumatic stress disorder (PTSD) is a psychiatric illness that can develop after having experienced traumatic, often life treathening, events. The symptoms often leads to significant subjective suffering, and may limit vocational and social functioning.

Intensive trauma treatment with Eye Movement Desensitization and Reprocessing (EMDR) and Prolonged Exposure (PE) of patients with PTSD has not previously been conducted in an inpatient setting in Norway. In this study we foremost seek to examine if this combined intervention, given at a five day inpatient unit, is suitable to a norwegian PTSD population and clinical setting. We will do this by systematically gathering information about how many drop out of the treatment program, and if so, at what stage of the program. We will also ask the patients to complete a short questionnaire about how they viewed the treatment program overall, and the separate parts of the program. We also wish to examine how the patients experienced the intervention, and in what way it contributet to their possible improvemen,t through a qualitative interview. We will also use well established clinical self report questionnaires to investigate if the patients who participate in the treatment program will experience an improvement of their PTSD symptoms and improved functioning, and examine if this possible improvement lasts two and six months post treament.

Method: This is a pilotstudy where a total of twelve patients with PTSD will be recruited from the Nydalen outpatient department, Oslo University Hospital. The patients have to satisfy the studies inclusion criteria, including having experienced at least two traumatic experiences, and had at least one previous psyhotherapeutic treament. The patients will be examined with validated self report questionnaires before and after the intervention, as well as after two and six months post treatment. Six patients will be invited to participate in a qualitative interview focusing on their experience of the intervention.

The Intervention: Treatment program monday to friday with daily PE and EMDR sessions, physical activity between sessions, in vivo exposure treament and psychoeducational groups. Daily rotation of both EMDR and PE therapists. Multidisiplinary team attached to each patient.

Significance of the study: Intensive inpatient trauma treatment with EMDR and PE have not previously been done in Norway. It has neither, as far as we know, been conducted any qualitative studies of this intensive combined treatment method internationally.The project wish to contribute to change trauma treatment in our hospital from a stabilisation focus to a focus on active trauma processing and treatment, to increase our staffs and therapists competency in trauma treatment, and to further the national and international body of knowledge about how patients with PTSD best can experience functional and symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Satisfying diagnostic criteria for PTSD (based on the MINI diagnostic interview)
* having experienced at least two traumatic experiences
* had at least one previous psyhotherapeutic treament (> 3 months)
* ability to speak a scandinacian language,

Exclusion Criteria:

* IQ <70, substance abuse
* regular use of benzodiazapines
* serious suicidality (suicide attempt last 3 months)
* neurological illness or significant headinjury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
PTSD symptom reduction | 2 weeks, 2 months, 6 months
  Change on Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) questionnaire. Max score 80, minimum score 0. 0= no PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Julie Evensen, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaage-Kowalzik V, Engeset J, Jakobsen M, Evensen JH. "The world does not look the same anymore": The experiences of patients six months after finishing an intensive trauma treatment program. BMC Psychol. 2025 Dec 12;14(1):77. doi: 10.1186/s40359-025-03826-2. PMID 41382171
- [Derived] Vaage-Kowalzik V, Engeset J, Jakobsen M, Evensen JH. Educational, but demanding: the experience of therapists in an intensive inpatient trauma treatment program. Front Psychol. 2025 Aug 29;16:1581055. doi: 10.3389/fpsyg.2025.1581055. eCollection 2025. PMID 40949339
- [Derived] Vaage-Kowalzik V, Engeset J, Jakobsen M, Andreassen W, Evensen JH. Exhausting, but necessary: the lived experience of participants in an intensive inpatient trauma treatment program. Front Psychol. 2024 May 28;15:1341716. doi: 10.3389/fpsyg.2024.1341716. eCollection 2024. PMID 38863672